CLINICAL TRIAL: NCT00122421
Title: The Impact of Pharmacist Recommendations on Quality of Care in Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Rebecca J. Cunningham, MD, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2003-P-000950/2; BWH
Record Dates: First submitted 2005-07-19; First posted 2005-07-22 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; quality of care; pharmacist recommendations
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- pharmacist recommendation (Active Comparator): recommendations based on chart review by pharmacist, given to pcp at time of visit
  Interventions: Behavioral: Pharmacist recommendations to primary care providers; Other: pharmacist recommendations
- usual care (No Intervention): usual care

INTERVENTIONS:
Behavioral: Pharmacist recommendations to primary care providers — recommendations based on chart review by pharmacist, given to pcp at time of visit
  Arms: pharmacist recommendation
Other: pharmacist recommendations — recommendations based on chart review by pharmacist, given to pcp at time of visit
  Arms: pharmacist recommendation

SUMMARY:
The goal of this study is to investigate a comprehensive provider-focused intervention to improve the quality of care for diabetic patients in a large primary care practice at Brigham and Women's Hospital. This will be accomplished through pharmacist recommendations provided to primary care providers prior to routine scheduled office visits for diabetic patients.

DETAILED DESCRIPTION:
Type II diabetes mellitus is an increasingly common condition among adults in the United States and is associated with substantial morbidity and mortality. The microvascular and macrovascular complications of diabetes lead to significant disability and early mortality, in addition to tremendous costs to the healthcare system. It has been clearly demonstrated, that both microvascular and macrovascular complications can be reduced through specific interventions that can be carried out by office-based primary care physicians. Despite the accumulation of evidence regarding specific interventions that can reduce diabetes-related morbidity and mortality, multiple studies have shown that the care provided for diabetic patients frequently falls short of recommended standards.

The researcher's goal is to investigate a comprehensive, provider-focused intervention to improve the quality of care for diabetic patients in a large, primary care practice at Brigham and Women's Hospital. This will be accomplished through pharmacist-delivered recommendations provided to primary care providers prior to routine scheduled office visits for diabetic patients.

Adult diabetic patients age 18 years and older receiving primary care in the Brigham Internal Medicine Associates (BIMA) practice will be randomized to intervention and control groups, based on the practice subset (Suite) within BIMA in which they receive their ongoing care. Patients who receive care from providers in Suites A, B, E, and F will be assigned to the intervention group, while patients who receive care from providers in Suites C, D, G, and H will be assigned to the control group. Patients will not be contacted regarding the study; providers who practice in the intervention Suites will receive specific written recommendations regarding optimal diabetes care parameters from our study pharmacist prior to each patient's visit. Providers who practice in the control Suites will not be contacted. Pre- and post-intervention compliance with multiple diabetes quality-of-care measures (eg, Hemoglobin A1c measurement, LDL cholesterol measurement, pneumococcal vaccination, etc.) will be assessed in the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of diabetes
* Age 18 years or older
* Identifiable primary care physician (PCP)
* Attendance at index appointment with PCP

Exclusion Criteria:

* No assigned PCP
* Non-attendance at PCP appointment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2003-06; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Compliance with process measures at 30 days after the index primary care visit | 30 days
  aspirin use, ace inhibitor use, a1c measurement

SECONDARY OUTCOMES:
Percentage of pharmacist recommendations accepted by primary care providers within 30 days after index visit | 30 days
  %adherence to recommendations

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca J Cunningham, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States